CLINICAL TRIAL: NCT00143949
Title: Renin Angiotensin System Blockage-DN (RASS)
Brief Title: Renin Angiotensin System Study (RASS/B-RASS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Mauer, MD (Individual)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Merck Sharp & Dohme LLC (Industry); Merck Frosst Canada Ltd. (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Organization: University of Minnesota (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 9601M10705
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; nephropathy; kidney; retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Kidney Diseases; Retinal Diseases | interventions — Enalapril; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: enalapril
Drug: losartan

SUMMARY:
To determine if renin angiotensin medications can prevent or delay the onset of diabetic kidney disease.

DETAILED DESCRIPTION:
The primary objective of this research is to determine, in type 1 (insulin-dependent) diabetic patients without hypertension, diabetic nephropathy (DN), or levels of microalbuminuria (MA) predictive of underlying, already established serious lesion of diabetic nephropathy, if inhibition of renin-angiotensin system (RAS) activity can prevent or retard the rate of development of the histologic lesions associated with DN. This primary prevention study is designed to examine the effect of pharmacologic intervention on the earliest stages of diabetic kidney disease. At the stage of overt DN intervention studies have shown only a slowing, as opposed to arrest, in disease progression, and benefit a minority of treated patients. At the MA stage the renal lesions of DN are already usually firmly established; moreover, progression in MA patients may occur despite strict glycemic or anti-hypertensive control. Renal histologic change over time has been selected as the primary endpoint in order to study the early stages of this disease, since the time to functional endpoints from these earlier stages precludes practical study design.

Specific Aim 1 To recruit 285 type 1 diabetic patients who do not have hypertension, diabetic nephropathy, or predictive levels of microalbuminuria into a 5-year study to determine the effect of inhibition of renin-angiotensin system activity with either losartan (angiotensin II blocker) or enalapril (converting enzyme inhibitor) on the development of diabetic renal disease. This aim has been accomplished and the study is entitled the Renin-Angiotension System Study (RASS).

Specific Aim 2 To obtain two percutaneous renal biopsies from each patient, the first, at entry into the study, and the second after five years of drug therapy with either losartan or enalapril.

Hypothesis Reduction of renin-angiotensin system activity will prevent or retard the development of histologic change in the kidney associated with diabetic nephropathy.

A secondary objective of this study is to evaluate retinal lesions in the RASS cohort of patients in order to determine the relationship of these findings to the histologic changes of DN and to examine the effects of RAS inhibition and/or systemic blood pressure (BP) on the development and progression of diabetic retinopathy. This ancillary study has the following aims:

Specific Aim To obtain baseline, 2.5 and 5 year retinal fundus photographs in the RASS patients.

Hypothesis Cross-sectional and longitudinal relationships of retinal and renal structural abnormalities will emerge which will improve the predictive value of renal functional tests. Reduction of rennin-angiotensin system activity will prevent or retard the development of diabetic retinal lesions

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetic (DM) for 2-20 yrs
* type 1 DM onset prior to 45; if onset was between ages 31-41, BMI <26; onset 41-45, positive GAD or ICA required
* normal or increased GFR
* normal BP
* normoalbuminuric (<20 ug/min on 2 of 3 time overnight urine collections)

Exclusion Criteria:

* type 1 DM duration longer than 20 yrs
* hypertension (>85/135 mmHg)
* reduced GFR (<90 ml/min/1.73m2)
* microalbuminuria
* solitary kidney or evidence of unilateral renal disease
* evidence of other important kidney disease by history, ultrasound or biopsy
* other chronic diseases or conditions such as cystic fibrosis, serious mental illness, severe mental retardation, etc.
* pregnancy or females planning pregnancy within 2 years were excluded due to the drugs being used
* compliance (pt not taking at least 85% of two week placebo were excluded)

Ages: 16 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 285 (Actual)
Dates: Start 1997-03; Primary Completion 2007-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To recruit 285 type 1 DM Pts without HTN, diabetic nephropathy, or microalbuminuria into a 5-year study to determine the effect of inhibition RAS with either losartan or enalapril. | 5 year
To obtain two percutaneous renal biopsies from each patient, five years apart. | 5 year

SECONDARY OUTCOMES:
To evaluate retinal lesions in RASS cohort to determine relationship to the histologic changes of DN and the effects of RAS inhibition and/or systemic blood pressure. | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: S M Mauer, MD, Principal Investigator — University of Minnesota
Locations (3):
- Canada (3):
  - Mt Sinai Hospital, University of Toronto (Clinical Ctr), Toronto, Ontario
  - Royal Victoria Hospital, McGill University (Data Center), Montreal, Quebec
  - Montreal Childrens Hospital, McGill University (Clinical Ctr), Montreal, Quebec

REFERENCES:
- [Background] Mauer M, Zinman B, Gardiner R, Drummond KN, Suissa S, Donnelly SM, Strand TD, Kramer MS, Klein R, Sinaiko AR. ACE-I and ARBs in early diabetic nephropathy. J Renin Angiotensin Aldosterone Syst. 2002 Dec;3(4):262-9. doi: 10.3317/jraas.2002.048. PMID 12584670
- [Derived] Limonte CP, Prince DK, Hoofnagle AN, Galecki A, Hirsch IB, Tian F, Waikar SS, Looker HC, Nelson RG, Doria A, Mauer M, Kestenbaum BR, de Boer IH. Associations of Biomarkers of Tubular Injury and Inflammation with Biopsy Features in Type 1 Diabetes. Clin J Am Soc Nephrol. 2024 Jan 1;19(1):44-55. doi: 10.2215/CJN.0000000000000333. Epub 2023 Oct 23. PMID 37871959
- [Derived] Robiner WN, Strand TD, Mauer M; Renin Angiotensin System Study (RASS) Group. Adherence and renal biopsy feasibility in the Renin Angiotensin-System Study (RASS) primary prevention diabetes trial. Diabetes Res Clin Pract. 2013 Oct;102(1):25-34. doi: 10.1016/j.diabres.2013.06.004. Epub 2013 Sep 17. PMID 24050942
- [Derived] Harindhanavudhi T, Mauer M, Klein R, Zinman B, Sinaiko A, Caramori ML; Renin Angiotensin System Study (RASS) group. Benefits of Renin-Angiotensin blockade on retinopathy in type 1 diabetes vary with glycemic control. Diabetes Care. 2011 Aug;34(8):1838-42. doi: 10.2337/dc11-0476. Epub 2011 Jun 29. PMID 21715517
- [Derived] Klein R, Myers CE, Klein BE, Zinman B, Gardiner R, Suissa S, Sinaiko AR, Donnelly SM, Goodyer P, Strand T, Mauer M. Relationship of blood pressure to retinal vessel diameter in type 1 diabetes mellitus. Arch Ophthalmol. 2010 Feb;128(2):198-205. doi: 10.1001/archophthalmol.2009.391. PMID 20142543
- [Derived] Mauer M, Zinman B, Gardiner R, Suissa S, Sinaiko A, Strand T, Drummond K, Donnelly S, Goodyer P, Gubler MC, Klein R. Renal and retinal effects of enalapril and losartan in type 1 diabetes. N Engl J Med. 2009 Jul 2;361(1):40-51. doi: 10.1056/NEJMoa0808400. PMID 19571282